CLINICAL TRIAL: NCT03963739
Title: Influence of Primary Treatment for Prostate Cancer on Work Experience (PCW)
Brief Title: Effect of Treatment on Work Experience in Patients With Stage I-III Prostate Cancer
Acronym: PCW
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00056621; NCI-2018-03915 (Registry Identifier: NCI Trial Identifier); P30CA012197 (NIH); UG1CA189824 (NIH); NCI-2018-03915 (Registry Identifier: NCI CTRP); WF-1802 (Other: WF NCORP RB)
Record Dates: First submitted 2019-05-21; First posted 2019-05-28 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Prostate Adenocarcinoma; Stage I Prostate Cancer; Stage II Prostate Cancer; Stage III Prostate Cancer
Keywords: Prostate; Adenocarcinoma
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Race: Non-Hispanic African American: Patients undergo an interview over 40-60 minutes at baseline and 3 and 6 months after treatment to describe and compare changes in ability to work and employment status/income.
  Interventions: Other: Interview; Other: Questionnaire Administration
- Race: Non-Hispanic White: Patients undergo an interview over 40-60 minutes at baseline and 3 and 6 months after treatment to describe and compare changes in ability to work and employment status/income.
  Interventions: Other: Interview; Other: Questionnaire Administration
- Income: Lower Income: Patients undergo an interview over 40-60 minutes at baseline and 3 and 6 months after treatment to describe and compare changes in ability to work and employment status/income.
  Interventions: Other: Interview; Other: Questionnaire Administration
- Income: Higher Income: Patients undergo an interview over 40-60 minutes at baseline and 3 and 6 months after treatment to describe and compare changes in ability to work and employment status/income.
  Interventions: Other: Interview; Other: Questionnaire Administration

INTERVENTIONS:
Other: Interview — Undergo interview
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
The objective of this study is to examine how adenocarcinoma of the prostate treatment differentially affects African American men's ability to work and to describe and compare changes in work ability (as measured through self-reported global work ability item) reported by African American and white adenocarcinoma of the prostate survivors before treatment and 6 months after treatment completion.

DETAILED DESCRIPTION:
This observational, longitudinal study will recruit approximately 255 patients through the Wake Forest National Cancer Institute Community Oncology Research Program (NCORP) Research Base (WF NCORP RB). The recruitment goal will be to have 160 participants who complete the interviewer-administered Structured Questionnaire at all three time points. All participants will be administered the first Structured Questionnaire prior to a prostatectomy or initiation of radiation therapy to treat adenocarcinoma of the prostate. Participants will also be administered Structured Questionnaires at three and six months after the prostatectomy or completion of radiation therapy. For most patients, the time between study enrollment and completion of participation will be approximately 6 - 10 months. Interviewer-administered Structured Questionnaires will address work ability, job characteristics, presence of symptoms associated with adenocarcinoma of the prostate treatment, and general background information.

ELIGIBILITY:
Inclusion Criteria:

* Male diagnosed with adenocarcinoma of the prostate, stage I, II, or III. Patient may have already received hormonal therapy or expect to receive hormonal therapy as treatment for adenocarcinoma of the prostate
* Scheduled to undergo prostatectomy or initiate radiation for primary curative treatment of adenocarcinoma of the prostate within 90 days of enrollment
* Self-identify as African American/black, non-Hispanic OR white, non-Hispanic; Participants are considered African American for recruitment purposes if they (1) identify solely as African American for race OR (2) identify as African American and white for race, but do not identify as also being of another race. Participants are considered white for recruitment purposes if they select white and no other race. (These identities are based on participant self-report during the screening process.)
* Eastern Cooperative Oncology Group (ECOG) score = 0 or 1
* Worked within the past 14 days prior to screening (no minimum number of hours required) OR (a) worked at some point between March 1, 2020 - March 14, 2020 and (b) subsequently lost job involuntarily due to COVID-19.
* Intends to be working 6 months from screening (if opportunity to work is available pending the COVID-19 pandemic considerations)
* Patient is willing to provide answers on the patient eligibility questionnaire regarding household income
* Age at time of screening is > or = 18
* Can speak and understand spoken English
* Ability to understand an informed consent document (even if only verbally) and willingness to agree to informed consent document
* Access to telephone or willingness to travel to National Cancer Institute (NCI) Community Oncology Research Program (NCORP) site for each of the three interviewer-administered structured questionnaires
* Able to hear sufficiently to understand a conversation determined by a simple test given at screening
* Has not previously had a prostatectomy, radiation therapy, or chemotherapy to treat adenocarcinoma of the prostate
* Not expected (at time of screening) to receive chemotherapy for primary treatment of adenocarcinoma of the prostate

Exclusion Criteria:

* Patient has received therapy for any other cancer within last 3 years (except for non-melanoma skin cancer)
* Patient plans to receive therapy for any other cancer within the next year (except for non-melanoma skin cancer)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosed with adenocarcinoma of the prostate, stage I, II, or III and scheduled to undergo prostatectomy or initiate radiation
Sampling Method: Non-Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2019-07-19 (Actual); Primary Completion 2025-03-25 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Change in work ability measured by Global Work Ability | Baseline up to 6 months after treatment completion
  Calculate 95% confidence intervals around the work ability score and the change in the work ability score. A two group t-test will be used to compare changes in the work ability score by race (white, African American), followed by a general linear model to compare changes in work ability with adjustment for demographic, work environment, and other baseline characteristics.

SECONDARY OUTCOMES:
Trajectory of change in work ability at 3 months measured by Global Work Ability | Baseline up to 3 months after treatment completion
  Measured by Global Work Ability. Quantify this change using means and 95% confidence intervals. In mixed models to account for the repeated measures over time, will model this change by race, income, and the interaction between race and income. Will also test for race by time and income by time interactions to compare the trajectories of change over time.
Trajectory of change in work ability at 6 months measured by Global Work Ability | Baseline up to 6 months after treatment completion
  In mixed models to account for the repeated measures over time, will model this change by race, income, and the interaction between race and income. Will also test for race by time and income by time interactions to compare the trajectories of change over time.
Trajectory of change in work ability at 3 months measured by Work Limitations Questionnaire (WLQ) | From baseline to 3 months after treatment completion
  Quantify this change using means and 95% confidence intervals. In mixed models to account for the repeated measures over time, will model this change by race, income, and the interaction between race and income. Will also test for race by time and income by time interactions to compare the trajectories of change over time.
Trajectory of change in work ability at 6 months measured by Work Limitations Questionnaire (WLQ) | Baseline up to 6 months after treatment completion
  Quantify this change using means and 95% confidence intervals. In mixed models to account for the repeated measures over time, will model this change by race, income, and the interaction between race and income. Will also test for race by time and income by time interactions to compare the trajectories of change over time.
Trajectory of change in work ability at 3 months measured by employment status | Baseline up to 3 months after treatment completion
  A random effects logistic regression model (if binary) or multinomial model (if more than 2 categories) for modeling employment status. Backwards model selection and Akaike information criterion (AIC) criteria will be utilized to identify the best model fit.
Trajectory of change in work ability at 6 months measured by employment status | Baseline up to 6 months after treatment completion
  A random effects logistic regression model (if binary) or multinomial model (if more than 2 categories) for modeling employment status. Backwards model selection and AIC criteria will be utilized to identify the best model fit.
Difference between preferred and actual length of leave | Up to 3 months after treatment completion
  Examine whether demographics, treatment, psychosocial and physical effects of treatment, and work environment factors impact (a) desired and (b) actual length of leave following treatment for adenocarcinoma of the prostate. Factors that are significant at an alpha level of 0.25 or less or have significant interactions will be entered into a general linear model.
Difference between preferred and actual length of leave | Up to 6 months after treatment completion
  Examine whether demographics, treatment, psychosocial and physical effects of treatment, and work environment factors impact (a) desired and (b) actual length of leave following treatment for adenocarcinoma of the prostate. Factors that are significant at an alpha level of 0.25 or less or have significant interactions will be entered into a general linear model.

OTHER OUTCOMES:
Effect of race and income on treatment-related function, work environment, and type of treatment | Up to 6 months after treatment completion
  Will use interactions to test moderation effects of race and income on the relationship between adenocarcinoma of the prostate treatment-related function (bladder, bowel, and hormonal function), work environment (e.g., work demands, workplace control, and social support), and type of treatment (surgery or radiation therapy, hormonal treatment) regarding outcomes of work limitations (as measured by the Work Limitations Questionnaire), Global Work Ability item, employment status, and preferred and actual length. Work ability, as measured through the WLQ and the Global Work Ability measures, and preferred versus actual length of time off work will be modeled as continuous variables in general linear models; employment status will be modeled as dichotomous (logistic regression) or in a multinomial model depending on the distribution of responses.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Lesser, MD, Study Chair — Wake Forest University Health Sciences
Locations (326):
- United States (325):
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Kaiser Permanente-Ontario, Ontario, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Saint Francis Cancer Center, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Beebe South Coastal Health Campus, Frankford, Delaware
  - Beebe Medical Center, Lewes, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Island Urology-Hilo, Hilo, Hawaii
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Cancer Center - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Hawaii Diagnostic Radiology Services LLC, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - The Queen's Medical Center - West Oahu, ‘Ewa Beach, Hawaii
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Reid Health, Richmond, Indiana
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Saint Luke's Hospital, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Trinity Regional Medical Center, Fort Dodge, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Our Lady of the Lake Physicians Group - Medical Oncology, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates, Baton Rouge, Louisiana
  - Our Lady of the Lake Medical Oncology, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Covington, Covington, Louisiana
  - Northshore Oncology Associates-Covington, Covington, Louisiana
  - Mary Bird Perkins Cancer Center - Houma, Houma, Louisiana
  - Terrebonne General Medical Center, Houma, Louisiana
  - LSU Healthcare Network / Metairie Multi-Specialty Clinic, Metairie, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Bronson Battle Creek, Battle Creek, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Ascension Borgess Cancer Center, Oshtemo, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Holy Name Hospital, Teaneck, New Jersey
  - Wake Forest University at Clemmons, Clemmons, North Carolina
  - Nash General Hospital, Rocky Mount, North Carolina
  - Wake Forest Baptist Health - Wilkes Medical Center, Wilkesboro, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford South University Medical Center, Fargo, North Dakota
  - Southpointe-Sanford Medical Center Fargo, Fargo, North Dakota
  - Sanford Medical Center Fargo, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Saint Elizabeth Boardman Hospital, Boardman, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC-Miami Valley Hospital North, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Columbus Oncology and Hematology Associates, Dublin, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Central Ohio Breast and Endocrine Surgery, Gahanna, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Mercy Health - Saint Vincent Hospital, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Mercy Health Sylvania Radiation Oncology Center, Toledo, Ohio
  - Dayton Physicians LLC-Upper Valley, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Saint Joseph's/Candler - Bluffton Campus, Bluffton, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - South Carolina Cancer Specialists PC, Hilton Head Island, South Carolina
  - The Radiation Oncology Center-Hilton Head/Bluffton, Hilton Head Island, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - North Grove Medical Park, Spartanburg, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Spartanburg Medical Center - Mary Black Campus, Spartanburg, South Carolina
  - MGC Hematology Oncology-Union, Union, South Carolina
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - VCU Massey Cancer Center at Hanover Medical Park, Mechanicsville, Virginia
  - Bon Secours Westchester Emergency Center, Midlothian, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours DePaul Medical Center, Norfolk, Virginia
  - Bon Secours Maryview Medical Center, Portsmouth, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Bon Secours Cancer Institute at Reynolds Crossing, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Bon Secours Health Center at Harbour View, Suffolk, Virginia
  - Saint Michael Cancer Center, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Valley Medical Center, Renton, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Westfields Hospital/Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Clinic Stevens Point Center, Stevens Point, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
- FHP Health Center-Guam, Tamuning, GU, Guam

IPD SHARING:
Plan to Share IPD: Yes
Wake Forest NCORP Research Base is committed to following the NIH Statement on Sharing Research Data (http://grants.nih.gov/grants/guide/notice-files/NOT-OD-03-032.html). As of July 2018, the WF NCORP RB signed an agreement with NCI to contribute de-identified data and data dictionaries from clinical trials conducted through our RB to the NCI NCTN/NCORP data archive within 6 months of primary and non-primary publications of phase II/III and phase III trials to https://nctn-data-archive.nci.nih.gov/. This will become the primary means for sharing raw data, and we will adhere to the guidelines spelled out in the NCTN/NCORP Data Archive Usage Guide. De-identified data from studies not covered by the agreement (e.g., phase II and observational studies) will be made available upon request. All data files will be de-identified. De-identification procedures will meet the HIPAA criteria as detailed in the Code of Federal Regulations, Part 45, Section 164.514.
Time Frame: 6 months after publication for a 2 year duration
Access Criteria: upon request to NCORP@wakehealth.edu